CLINICAL TRIAL: NCT07394361
Title: The Effect of Clinical Pilates Training on Fatigue, Emotional State, Functional Capacity, Sleep and Quality of Life in Women With Systemic Lupus Erythematosus
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Emir İbrahim IŞIK (Other)
Responsible Party: Sponsor-Investigator, Emir İbrahim IŞIK, Asst. Prof., Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLE_KP_01; CukurovaU (Other: CukurovaU)
Record Dates: First submitted 2025-04-24; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-04

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus; Clinical Pilates
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will participate in supervised clinical Pilates exercises. These exercises will be administered in the form of group sessions, which are to be held twice per week. In addition to the home exercise program, which is to be followed for a period of eight weeks.
  Interventions: Other: Clinical Pilates Training; Other: Home exercise program
- Control group (Active Comparator): The control group will be provided with a home exercise program. This program will consist of stretching, relaxation, and strengthening exercises, to be performed three days a week for a period of eight weeks.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Clinical Pilates Training — Warm-up (5 min) Segmental extremity movements Centering Roll down
  Pilates exercises (35 min) One leg stretch Double leg stretch Shoulder bridge Chest lift Hundreds Side band Arm opening Cobra Swimming Push-up
  Cool-down (5 min) Cat stretching Camel stretching Relaxation exercises
  Arms: Intervention group
Other: Home exercise program — This program will consist of stretching, relaxation, and strengthening exercises, to be performed three days a week for a period of eight weeks.

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic, autoimmune, inflammatory disease with the potential to affect any organ in the body. The most frequently affected anatomical regions include the skin, joints, pleura, pericardium, kidneys and the central nervous system.

All systemic conditions observed in SLE cause functional deficiencies in daily life, fatigue, anxiety and depression, pain, sleep quality disorders, cognitive effects, cosmetic problems, social isolation, and all these characteristics negatively affect the quality of life of an individual with SLE.

The aim of this study is to investigate the effects of clinical pilates exercises on pain, fatigue, functional capacity, flexibility, emotional state, sleep and quality of life in patients with SLE.

DETAILED DESCRIPTION:
The Effect of Clinical Pilates Training on Fatigue, Emotional State, Functional Capacity, Sleep and Quality of Life in Women with Systemic Lupus Erythematosus

Systemic lupus erythematosus (SLE) is a chronic, autoimmune, inflammatory disease with the potential to affect any organ in the body. The most frequently affected anatomical regions include the skin, joints, pleura, pericardium, kidneys and the central nervous system.

All systemic conditions observed in SLE cause functional deficiencies in daily life, fatigue, anxiety and depression, pain, sleep quality disorders, cognitive effects, cosmetic problems, social isolation, and all these characteristics negatively affect the quality of life of an individual with SLE.

The aim of this study is to investigate the effects of clinical pilates exercises on pain, fatigue, functional capacity, flexibility, emotional state, sleep and quality of life in patients with SLE.

The objectives of this study are as follows:

1. To examine the effect of a home exercise program on physical and psychological parameters in patients with SLE.
2. To examine the effect of Pilates exercises to be performed under supervision added to the home exercise program on physical and psychological parameters in patients with SLE.
3. To evaluate the cost-effectiveness of a home exercise program and clinical Pilates exercises.

MATERIAL AND METHOD Criteria for inclusion in the study: being a woman between the 18 Years to 65 Years , meeting the American College of Rheumatology SLE diagnostic criteria, having low disease activity (SLEDAI ≤4), agreeing to participate in the study Exclusion criteria from the study: presence of malignancy, pregnancy, change of treatment within the last 3 months, use of steroids equivalent to >16 mg prednisolone for the last 3 months, have other rheumatic diseases, have a regular exercise habit (physical activity more than two times a week), have a disease that restricts physical activity (such as neurological disorder, orthopedic disorder, cognitive disorder, immobility), have serious heart, lung or kidney involvement, uncontrolled hypertension, severe anemia (hb <8 g/dL), having undergone orthopedic surgery in the last 6 months.

Following the provision of informed consent, participants will be randomly divided into two groups using a computer program. In addition to the home exercise program, which is to be followed for a period of eight weeks, the intervention group will participate in supervised clinical Pilates exercises. These exercises will be administered in the form of group sessions, which are to be held twice per week. The control group will be provided with a home exercise program. This program will consist of stretching, relaxation, and strengthening exercises, to be performed three days a week for a period of eight weeks.

Participants will be contacted by phone weekly to encourage compliance with the exercise regimen. In addition, participants will be given an exercise diary and instructed to record their exercise days in a systematic way. Participants who show less than 80% compliance with the exercise program during subsequent follow-ups will be excluded from the study. Patients enrolled in the study will undergo three evaluations. The first evaluation will be performed before the treatment and the second evaluation will be performed after the treatment. The third evaluation will be performed 3 months after the end of the treatment. Demographic information such as age, height, weight, body mass index, medications used and duration of illness will be documented before the intervention. The patient's pain during rest and activity will be evaluated using the visual analog scale (VAS). The patient's fatigue status will be evaluated using the fatigue severity scale (FSS). The emotional state of the patient will be evaluated using the hospital anxiety and depression scale (HADS). The functional capacity of the patient will be evaluated using a 6-minute walking test and a 30-second sitting test. The patient's flexibility will be evaluated using the sitting access test. The patient's hand grip strength will be evaluated using a hand dynamometer. The patient's sleep quality will be evaluated using the Jenkins sleep scale (JSS). The quality of life of the patient will be evaluated using the systemic lupus erythematosus quality of life scale (SLEQoL). The functional status of the patient will be evaluated using the health assessment questionnaire (HAQ).

ELIGIBILITY:
Inclusion Criteria:

* being a woman between the 18 Years to 65 Years ,
* meeting the American College of Rheumatology SLE diagnostic criteria,
* having low disease activity (SLEDAI ≤4),
* agreeing to participate in the study

Exclusion Criteria:

* presence of malignancy, pregnancy, change of treatment within the last 3 months,
* use of steroids equivalent to >16 mg prednisolone for the last 3 months, - -
* have other rheumatic diseases,
* have a regular exercise habit (physical activity more than two times a week),
* have a disease that restricts physical activity (such as neurological disorder, orthopedic disorder, cognitive disorder, immobility),
* have serious heart, lung or kidney involvement,
* uncontrolled hypertension,
* severe anemia (hb <8 g/dL),
* having undergone orthopedic surgery in the last 6 months

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female participants will be included to the study.
Enrollment: 30 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Fatigue status (Fatigue Severity Scale) | 5 months
  The patient's fatigue status will be evaluated using the fatigue severity scale (FSS). The FSS is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Grading of each item ranges from 1 to 7, where 1 indicates strong disagreement and 7 strong agreement, and the final score represents the mean value of the 9 items.

SECONDARY OUTCOMES:
Pain score (Visual Analog Scale) | 5 months
  The patient's pain during rest and activity will be evaluated using the visual analog scale (VAS). The visual analogue scale is a psychometric response scale that can be used in questionnaires. It is a measurement tool for subjective characteristics or attitudes that cannot be measured directly. When responding to a VAS item, respondents indicate their level of agreement with a statement by indicating a position along a continuous line between two endpoints.
Emotional state (Hospital Anxiety and Depression Scale) | 5 months
  The emotional state of the patient will be evaluated using the hospital anxiety and depression scale (HADS).
Functional capacity (6-minute walking test, 30-second sitting test, Handgrip measurement) | 5 months
  The functional capacity of the patient will be evaluated using a 6-minute walking test and a 30-second sitting test. The patient's flexibility will be evaluated using the sitting access test. The patient's hand grip strength will be evaluated using a hand dynamometer.
Sleep quality (Jenkins sleep scale) | 5 months
  The patient's sleep quality will be evaluated using the Jenkins sleep scale (JSS).
SLE quality of life (Systemic lupus erythematosus quality of life scale) | 5 months
  The quality of life of the patient will be evaluated using the systemic lupus erythematosus quality of life scale (SLEQoL). SLEQoL is a lupus-specific scale developed in the United Kingdom. It is based on patient needs and the ability of patients to meet their needs. It is a simple questionnaire consisting of 25 items related to symptoms, functioning and disease-related issues. A 'correct' answer to the questions is considered 1 point and an 'incorrect' answer is considered 0 point. The total score is between 0 and 25, with a higher score indicating a lower quality of life.
Functional status (Health assessment questionnaire) | 5 months
  The functional status of the patient will be evaluated using the health assessment questionnaire (HAQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hashemi, S., Farahbakhsh, S., Fallahi, A., Daryanoosh, F., Babaei Beigi, M. A., & Jamshidian Tehrani, N. (2024). Aerobic and Anaerobic Exercise Benefits for Lupus: Fatigue, Fitness, and Life Quality. Iranian Rehabilitation Journal, 22(3), 499-508.
- [Result] Ismail AMA, Saad AE, Abd-Elrahman NAF, Elfahl AMA. Response of Lipid Profile to Laser Acupuncture along with Diet and Pilates Exercise in Obese Women with Systemic Lupus Erythematosus: a Randomized Controlled Trial. J Acupunct Meridian Stud. 2023 Aug 31;16(4):152-158. doi: 10.51507/j.jams.2023.16.4.152. PMID 37609770